CLINICAL TRIAL: NCT00185783
Title: Pilot Study of White Blood Cell Gene Expression in Critically Ill Patients With Severe Sepsis and Relative Adrenal Insufficiency After Hydrocortisone Administration
Brief Title: Impact of Hydrocortisone Administration on White Blood Cell Gene Expression in Patients With Severe Sepsis
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: University of Toronto (Other); University of Colorado, Denver (Other)
Responsible Party: Andrew J. Patterson, M.D., Ph.D., Stanford University
Other Study IDs: 95230; Stanford IRB Number 4593; Other Grant (Other Grant/Funding Number: Stanford University Department of Anesthesia)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Sepsis; Relative Adrenal Insufficiency
Keywords: Sepsis; Adrenal Insufficiency; Hydrocortisone; Gene Expression; Microarray; RNA; Critically Ill
MeSH Terms: conditions — Sepsis; Adrenal Insufficiency; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Hydrocortisone Administration (Standard of Care Therapy)

SUMMARY:
The purpose of this pilot study is to (1) examine the changes in gene expression in patients who suffer from severe sepsis and whose shock (inadequate oxygen delivery to vital organs) state does not respond to fluid and vasopressor administration, (2) to show that our sampling method of isolating RNA provides reliable and consistent data, (3) provide a basis for future gene expression studies in critically ill patients

DETAILED DESCRIPTION:
Severe sepsis is characterized by inadequate perfusion of vital organs due to infection. More than 750,000 cases of severe sepsis occur each year in the United States. Mortality among patients with severe sepsis ranges from 7% to 50%. Initiation of antibiotic therapy within the first hour of diagnosis as well as fluid resuscitation and hemodynamic stabilization are primary goals of therapy.

Steroid administration has been shown to improve outcome in the subset of severe sepsis patients suffering from relative adrenal insufficiency. Although initial studies using high dose short course steroid therapy did not demonstrate efficacy, more recent studies of low dose longer duration hydrocortisone administration demonstrated a significant reduction in mortality at 28 days. The mechanism by which steroid administration affords protection is unclear. We hypothesize that steroid administration changes white blood cell gene and protein expression in severe sepsis patients from an immuno-inflammatory profile to a pattern consistent with healing.

Our first specific aim is to obtain plasma and total cellular RNA from leukocytes in the blood of ten patients admitted to Stanford Medical Center with the diagnosis of severe sepsis and adrenal insufficiency. Significant and distinct variations in whole blood leukocyte gene expression patterns occur depending upon the method of RNA isolation. We will attempt to demonstrate that our sampling method provides reliable and consistent data.

Our second specific aim is to begin an analysis of gene expression patterns in white blood cells before and after steroid administration in patients suffering from severe sepsis with relative adrenal insufficiency. We will use a protocol for assessment of gene expression that was developed by members of our research team.

ELIGIBILITY:
Inclusion Criteria:

* Admission Diagnosis of Sepsis
* Evidence of Relative Adrenal Insufficiency
* Hypotension (Mean Arterial Pressure less than 60 mm Hg) Refractory to a. Fluid Resuscitation b. Dopamine infusion (greater than 5 micrograms/kg/min) c. Phenylephrine infusion (greater than 1 microgram/kg/min)

Exclusion Criteria:

* Use of Immunosuppressant Medications
* Immune Compromised Due to Disease (e.g., HIV infection)
* Transfusion of Blood Products within the past 7 Days
* Use of Cytokine Therapy (i.e., G-CSF)
* History of Bone Marrow Transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Stanford Hospital ICU with Sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2005-03; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Patterson, M.D., Ph.D., Principal Investigator — Stanford University, Dept. of Anesthesia, Division of Critical Care Medicine; Ann Weinacker, M.D.,, Principal Investigator — Stanford University, Dept. of Medicine, Div. of Pulmonary and Critical Care Medicine
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

REFERENCES:
- [Background] Spiegelman JI, Mindrinos MN, Oefner PJ. High-accuracy DNA sequence variation screening by DHPLC. Biotechniques. 2000 Nov;29(5):1084-90, 1092. doi: 10.2144/00295rr04. PMID 11084871
- [Background] Steinmetz LM, Mindrinos M, Oefner PJ. Combining genome sequences and new technologies for dissecting the genetics of complex phenotypes. Trends Plant Sci. 2000 Sep;5(9):397-401. doi: 10.1016/s1360-1385(00)01724-6. No abstract available. PMID 10973096
- [Background] Wang QT, Piotrowska K, Ciemerych MA, Milenkovic L, Scott MP, Davis RW, Zernicka-Goetz M. A genome-wide study of gene activity reveals developmental signaling pathways in the preimplantation mouse embryo. Dev Cell. 2004 Jan;6(1):133-44. doi: 10.1016/s1534-5807(03)00404-0. PMID 14723853
- [Background] Dellinger RP, Carlet JM, Masur H, Gerlach H, Calandra T, Cohen J, Gea-Banacloche J, Keh D, Marshall JC, Parker MM, Ramsay G, Zimmerman JL, Vincent JL, Levy MM; Surviving Sepsis Campaign Management Guidelines Committee. Surviving Sepsis Campaign guidelines for management of severe sepsis and septic shock. Crit Care Med. 2004 Mar;32(3):858-73. doi: 10.1097/01.ccm.0000117317.18092.e4. PMID 15090974
- [Background] Dellinger RP, Carlet JM, Masur H, Gerlach H, Calandra T, Cohen J, Gea-Banacloche J, Keh D, Marshall JC, Parker MM, Ramsay G, Zimmerman JL, Vincent JL, Levy MM. Surviving Sepsis Campaign guidelines for management of severe sepsis and septic shock. Intensive Care Med. 2004 Apr;30(4):536-55. doi: 10.1007/s00134-004-2210-z. Epub 2004 Mar 3. PMID 14997291
- [Background] Dellinger RP. Cardiovascular management of septic shock. Crit Care Med. 2003 Mar;31(3):946-55. doi: 10.1097/01.CCM.0000057403.73299.A6. No abstract available. PMID 12627010
- [Background] Annane D, Sebille V, Charpentier C, Bollaert PE, Francois B, Korach JM, Capellier G, Cohen Y, Azoulay E, Troche G, Chaumet-Riffaud P, Bellissant E. Effect of treatment with low doses of hydrocortisone and fludrocortisone on mortality in patients with septic shock. JAMA. 2002 Aug 21;288(7):862-71. doi: 10.1001/jama.288.7.862. PMID 12186604